CLINICAL TRIAL: NCT03030625
Title: Dose Intensification With a Focal Boost to Dominant Intraprostatic Lesion Using Volumetric Modulated Arc Therapy /Image Guided Radiotherapy in Patients With Localized Prostate Cancer
Brief Title: VMAT for Dominant Intraprostatic Lesion
Acronym: CaP-VMAT-DIL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CaP-VMAT-DIL
Record Dates: First submitted 2017-01-12; First posted 2017-01-25 (Estimated); Results first posted 2023-05-24 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; VMAT; Dominant Intraprostatic Lesion; Intensity modulated radiotherapy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IGRT/VMAT focal therapy boost to DIL (Other): Localized prostate cancer (PCa) of intermediate and high risk according to NCCN criteria
  Interventions: Radiation: IGRT/VMAT focal therapy boost to DIL

INTERVENTIONS:
Radiation: IGRT/VMAT focal therapy boost to DIL — Image-guided/VMAT focal Intensification dose to intraprostatic dominant lesion in men with localized prostate cancer (PCa) of intermediate and high risk (criteria NCCN) eligible to receive radiotherapy

SUMMARY:
The aim of this study was to determine the efficacy and safety of the implementation of a program of " image-guided focal Intensification dose to intraprostatic dominant lesion " in men with localized prostate cancer (PCa) of intermediate and high risk (criteria NCCN) eligible to receive radiotherapy in the Department of Radiation Oncology of HUP (Hospital Universitario de La Princesa), within the established dose escalation protocol with intensity modulated image-guided radiotherapy (IMRT / IGRT).

DETAILED DESCRIPTION:
The aim of this study was to determine the efficacy and safety of the implementation of a program of " image-guided focal Intensification dose to intraprostatic dominant lesion " in men with localized prostate cancer (PCa) of intermediate and high risk (criteria NCCN) eligible to receive radiotherapy in the Department of Radiation Oncology of HUP (Hospital Universitario de La Princesa), within the established dose escalation protocol with intensity modulated image-guided radiotherapy (IMRT / IGRT).

ELIGIBILITY:
Inclusion Criteria:

* Male > 18 years old with histologic diagnostic of prostate adenocarcinoma
* Clinical stage cT2a-T3b N0-1 M0 (AJCC 7 th edition)
* PSA (prostate-specific antigen) < 100 ng/ml
* Gleason score 6-10
* Life expectancy > 5 years
* Patients who accept the radiotherapy treatment
* Patients provided written informed consent before participating in the trial

Exclusion Criteria:

* Transurethral resection of the prostate or prior prostate surgery
* Previous pelvic radiotherapy
* Urethral stenosis with or without prior dilations
* IPSS>15
* Rectal diverticuli or rectal vascular malformations
* Metastatic disease
* Severe psychiatric or medical conditions that could hamper both treatment and follow-up

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-03-13 (Actual); Primary Completion 2023-01-25 (Actual); Study Completion 2023-01-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario de la Princesa, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arrayeh E, Westphalen AC, Kurhanewicz J, Roach M 3rd, Jung AJ, Carroll PR, Coakley FV. Does local recurrence of prostate cancer after radiation therapy occur at the site of primary tumor? Results of a longitudinal MRI and MRSI study. Int J Radiat Oncol Biol Phys. 2012 Apr 1;82(5):e787-93. doi: 10.1016/j.ijrobp.2011.11.030. Epub 2012 Feb 11. PMID 22331003
- [Background] Cellini N, Morganti AG, Mattiucci GC, Valentini V, Leone M, Luzi S, Manfredi R, Dinapoli N, Digesu' C, Smaniotto D. Analysis of intraprostatic failures in patients treated with hormonal therapy and radiotherapy: implications for conformal therapy planning. Int J Radiat Oncol Biol Phys. 2002 Jul 1;53(3):595-9. doi: 10.1016/s0360-3016(02)02795-5. PMID 12062602
- [Background] Pucar D, Hricak H, Shukla-Dave A, Kuroiwa K, Drobnjak M, Eastham J, Scardino PT, Zelefsky MJ. Clinically significant prostate cancer local recurrence after radiation therapy occurs at the site of primary tumor: magnetic resonance imaging and step-section pathology evidence. Int J Radiat Oncol Biol Phys. 2007 Sep 1;69(1):62-9. doi: 10.1016/j.ijrobp.2007.03.065. PMID 17707266
- [Background] Mouraviev V, Villers A, Bostwick DG, Wheeler TM, Montironi R, Polascik TJ. Understanding the pathological features of focality, grade and tumour volume of early-stage prostate cancer as a foundation for parenchyma-sparing prostate cancer therapies: active surveillance and focal targeted therapy. BJU Int. 2011 Oct;108(7):1074-85. doi: 10.1111/j.1464-410X.2010.10039.x. Epub 2011 Apr 13. PMID 21489116
- [Background] Peeters ST, Heemsbergen WD, Koper PC, van Putten WL, Slot A, Dielwart MF, Bonfrer JM, Incrocci L, Lebesque JV. Dose-response in radiotherapy for localized prostate cancer: results of the Dutch multicenter randomized phase III trial comparing 68 Gy of radiotherapy with 78 Gy. J Clin Oncol. 2006 May 1;24(13):1990-6. doi: 10.1200/JCO.2005.05.2530. PMID 16648499
- [Background] Kuban DA, Tucker SL, Dong L, Starkschall G, Huang EH, Cheung MR, Lee AK, Pollack A. Long-term results of the M. D. Anderson randomized dose-escalation trial for prostate cancer. Int J Radiat Oncol Biol Phys. 2008 Jan 1;70(1):67-74. doi: 10.1016/j.ijrobp.2007.06.054. Epub 2007 Aug 31. PMID 17765406
- [Background] Beckendorf V, Guerif S, Le Prise E, Cosset JM, Bougnoux A, Chauvet B, Salem N, Chapet O, Bourdain S, Bachaud JM, Maingon P, Hannoun-Levi JM, Malissard L, Simon JM, Pommier P, Hay M, Dubray B, Lagrange JL, Luporsi E, Bey P. 70 Gy versus 80 Gy in localized prostate cancer: 5-year results of GETUG 06 randomized trial. Int J Radiat Oncol Biol Phys. 2011 Jul 15;80(4):1056-63. doi: 10.1016/j.ijrobp.2010.03.049. Epub 2010 Dec 14. PMID 21147514
- [Background] Dearnaley DP, Jovic G, Syndikus I, Khoo V, Cowan RA, Graham JD, Aird EG, Bottomley D, Huddart RA, Jose CC, Matthews JH, Millar JL, Murphy C, Russell JM, Scrase CD, Parmar MK, Sydes MR. Escalated-dose versus control-dose conformal radiotherapy for prostate cancer: long-term results from the MRC RT01 randomised controlled trial. Lancet Oncol. 2014 Apr;15(4):464-73. doi: 10.1016/S1470-2045(14)70040-3. Epub 2014 Feb 26. PMID 24581940
- [Background] Zietman AL, Bae K, Slater JD, Shipley WU, Efstathiou JA, Coen JJ, Bush DA, Lunt M, Spiegel DY, Skowronski R, Jabola BR, Rossi CJ. Randomized trial comparing conventional-dose with high-dose conformal radiation therapy in early-stage adenocarcinoma of the prostate: long-term results from proton radiation oncology group/american college of radiology 95-09. J Clin Oncol. 2010 Mar 1;28(7):1106-11. doi: 10.1200/JCO.2009.25.8475. Epub 2010 Feb 1. PMID 20124169
- [Background] Zapatero A, Garcia-Vicente F, Martin de Vidales C, Cruz Conde A, Ibanez Y, Fernandez I, Rabadan M. Long-term results after high-dose radiotherapy and adjuvant hormones in prostate cancer: how curable is high-risk disease? Int J Radiat Oncol Biol Phys. 2011 Dec 1;81(5):1279-85. doi: 10.1016/j.ijrobp.2010.07.1975. Epub 2010 Oct 6. PMID 20932659
- [Background] King CR, Fowler JF. A simple analytic derivation suggests that prostate cancer alpha/beta ratio is low. Int J Radiat Oncol Biol Phys. 2001 Sep 1;51(1):213-4. doi: 10.1016/s0360-3016(01)01651-0. No abstract available. PMID 11516871
- [Background] Turkbey B, Albert PS, Kurdziel K, Choyke PL. Imaging localized prostate cancer: current approaches and new developments. AJR Am J Roentgenol. 2009 Jun;192(6):1471-80. doi: 10.2214/AJR.09.2527. PMID 19457807
- [Background] Barentsz JO, Richenberg J, Clements R, Choyke P, Verma S, Villeirs G, Rouviere O, Logager V, Futterer JJ; European Society of Urogenital Radiology. ESUR prostate MR guidelines 2012. Eur Radiol. 2012 Apr;22(4):746-57. doi: 10.1007/s00330-011-2377-y. Epub 2012 Feb 10. PMID 22322308
- [Background] Ippolito E, Mantini G, Morganti AG, Mazzeo E, Padula GD, Digesu C, Cilla S, Frascino V, Luzi S, Massaccesi M, Macchia G, Deodato F, Mattiucci GC, Piermattei A, Cellini N. Intensity-modulated radiotherapy with simultaneous integrated boost to dominant intraprostatic lesion: preliminary report on toxicity. Am J Clin Oncol. 2012 Apr;35(2):158-62. doi: 10.1097/COC.0b013e318209cd8f. PMID 21336090
- [Background] Pinkawa M, Attieh C, Piroth MD, Holy R, Nussen S, Klotz J, Hawickhorst R, Schafer W, Eble MJ. Dose-escalation using intensity-modulated radiotherapy for prostate cancer--evaluation of the dose distribution with and without 18F-choline PET-CT detected simultaneous integrated boost. Radiother Oncol. 2009 Nov;93(2):213-9. doi: 10.1016/j.radonc.2009.07.014. Epub 2009 Aug 28. PMID 19717197
- [Background] Pinkawa M, Piroth MD, Holy R, Klotz J, Djukic V, Corral NE, Caffaro M, Winz OH, Krohn T, Mottaghy FM, Eble MJ. Dose-escalation using intensity-modulated radiotherapy for prostate cancer - evaluation of quality of life with and without (18)F-choline PET-CT detected simultaneous integrated boost. Radiat Oncol. 2012 Jan 30;7:14. doi: 10.1186/1748-717X-7-14. PMID 22289620
- [Background] Wong WW, Schild SE, Vora SA, Ezzell GA, Nguyen BD, Ram PC, Roarke MC. Image-guided radiotherapy for prostate cancer: a prospective trial of concomitant boost using indium-111-capromab pendetide (ProstaScint) imaging. Int J Radiat Oncol Biol Phys. 2011 Nov 15;81(4):e423-9. doi: 10.1016/j.ijrobp.2011.01.048. Epub 2011 Apr 7. PMID 21477947
- [Background] Ellis RJ, Zhou H, Kim EY, Fu P, Kaminsky DA, Sodee B, Colussi V, Vance WZ, Spirnak JP, Kim C, Resnick MI. Biochemical disease-free survival rates following definitive low-dose-rate prostate brachytherapy with dose escalation to biologic target volumes identified with SPECT/CT capromab pendetide. Brachytherapy. 2007 Jan-Mar;6(1):16-25. doi: 10.1016/j.brachy.2006.11.002. PMID 17284381
- [Background] Miralbell R, Molla M, Rouzaud M, Hidalgo A, Toscas JI, Lozano J, Sanz S, Ares C, Jorcano S, Linero D, Escude L. Hypofractionated boost to the dominant tumor region with intensity modulated stereotactic radiotherapy for prostate cancer: a sequential dose escalation pilot study. Int J Radiat Oncol Biol Phys. 2010 Sep 1;78(1):50-7. doi: 10.1016/j.ijrobp.2009.07.1689. Epub 2009 Nov 10. PMID 19910135
- [Background] Fonteyne V, Villeirs G, Speleers B, De Neve W, De Wagter C, Lumen N, De Meerleer G. Intensity-modulated radiotherapy as primary therapy for prostate cancer: report on acute toxicity after dose escalation with simultaneous integrated boost to intraprostatic lesion. Int J Radiat Oncol Biol Phys. 2008 Nov 1;72(3):799-807. doi: 10.1016/j.ijrobp.2008.01.040. Epub 2008 Apr 11. PMID 18407430
- [Background] De Meerleer G, Villeirs G, Bral S, Paelinck L, De Gersem W, Dekuyper P, De Neve W. The magnetic resonance detected intraprostatic lesion in prostate cancer: planning and delivery of intensity-modulated radiotherapy. Radiother Oncol. 2005 Jun;75(3):325-33. doi: 10.1016/j.radonc.2005.04.014. PMID 15967524
- [Background] Zelefsky MJ, Cohen G, Zakian KL, Dyke J, Koutcher JA, Hricak H, Schwartz L, Zaider M. Intraoperative conformal optimization for transperineal prostate implantation using magnetic resonance spectroscopic imaging. Cancer J. 2000 Jul-Aug;6(4):249-55. PMID 11038145
- [Background] Brenner DJ, Hall EJ. Fractionation and protraction for radiotherapy of prostate carcinoma. Int J Radiat Oncol Biol Phys. 1999 Mar 15;43(5):1095-101. doi: 10.1016/s0360-3016(98)00438-6. PMID 10192361
- [Background] Williams SG, Taylor JM, Liu N, Tra Y, Duchesne GM, Kestin LL, Martinez A, Pratt GR, Sandler H. Use of individual fraction size data from 3756 patients to directly determine the alpha/beta ratio of prostate cancer. Int J Radiat Oncol Biol Phys. 2007 May 1;68(1):24-33. doi: 10.1016/j.ijrobp.2006.12.036. PMID 17448868
- [Background] Vogelius IR, Bentzen SM. Meta-analysis of the alpha/beta ratio for prostate cancer in the presence of an overall time factor: bad news, good news, or no news? Int J Radiat Oncol Biol Phys. 2013 Jan 1;85(1):89-94. doi: 10.1016/j.ijrobp.2012.03.004. Epub 2012 May 30. PMID 22652106

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IGRT/VMAT Focal Therapy Boost to DIL
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | IGRT/VMAT Focal Therapy Boost to DIL
Number analyzed (Participants) | 30
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 72.0 [67.7 to 76.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 30
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Spain | 30
Clinical T stage [Count of Participants; unit: Participants] — Clinical stage assessed by TNM ajcc seventh edition considering T2 less invasive than T3
  Participants
    T2: Tumor confinent whitin prostate | 23
    T3: Tumor extends through the prostate capsule | 7
Gleason group (ISUP 2014/WHO 2016) [Count of Participants; unit: Participants] — Gleason group classification for prostate cancer were used considering Group 1 as less aggressive and Group 5 most aggressive
  Participants
    Group 1: | 6
    Group 2 | 13
    Group 3 | 7
    Group 4 | 2
    Group 5 | 2
Pre-treatment PSA (ng/ml) [Median (Inter-Quartile Range); unit: ng/ml] | 8.5 [5.5 to 14.5]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Biochemical Failure at 5 Years
Description: Biochemical failure determined according to the Phoenix definition (nadir PSA + 2 ng/ml)
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Groups:
- IGRT/VMAT Focal Therapy Boost to DIL: Localized prostate cancer (PCa) of intermediate and high risk according to NCCN criteria
  IGRT/VMAT focal therapy boost to DIL: Image-guided/VMAT focal Intensification dose to intraprostatic dominant lesion in men with localized prostate cancer (PCa) of intermediate and high risk (criteria NCCN) eligible to receive radiotherapy: 35 daily fractions of 2.17 Gy with a concomitant focal boost to the intraprostatic nodule of 2.43 Gy
Arm/Group | IGRT/VMAT Focal Therapy Boost to DIL
Number analyzed (Participants) | 30
Participants
  Yes | 0
  No | 30

2. Primary Outcome: Local Control
Description: An image complete response was defined as disappearance of all morphological and functional lesions in mpMRI 6 to 9 months after radiotherapy.
Time Frame: 6 and 9 months following radiotherapy
Measure: Count of Participants; unit: Participants
Arm/Group | IGRT/VMAT Focal Therapy Boost to DIL
Number analyzed (Participants) | 30
Participants
  Yes | 30
  No | 0

3. Primary Outcome: Acute and Late Rectal and Urinary Complications
Description: Acute and late rectal and urinary complications defined as the number of participants with treatment-related adverse events assessed by Common Terminology Criteria for Adverse Events CTCAE v4.0 and Radiation- Therapy Oncology Group/ European Organization for Research and Treatment of Cancer RTOG/EORTC scales (been 0: no toxicity and 4: most severe toxicity).
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | IGRT/VMAT Focal Therapy Boost to DIL
Number analyzed (Participants) | 30
Participants
  Acute rectal: Grade 0 | 28
  Acute rectal: Grade 1 | 2
  Acute rectal: Grade 2 | 0
  Acute rectal: Grade >2 | 0
  Acute urinary: Grade 0 | 11
  Acute urinary: Grade 1 | 13
  Acute urinary: Grade 2 | 6
  Acute urinary: Grade >2 | 0
  Late rectal: Grade 0 | 27
  Late rectal: Grade 1 | 3
  Late rectal: Grade 2 | 0
  Late rectal: Grade >2 | 0
  Late urinary: Grade 0 | 27
  Late urinary: Grade 1 | 3
  Late urinary: Grade 2 | 0
  Late urinary: Grade >2 | 0

4. Secondary Outcome: Number of Participants Free of Biochemical Progression
Description: Biochemical disease-free survival according to the Phoenix definition (PSA >2 ng/mL above the currently observed PSA nadir. Defined as the time from enrollment to progression of biochemical disease, or death from any cause, or censoring at the date of the last contact.
Time Frame: 5 years
Population: Localized prostate cancer (PCa) of intermediate and high risk
Measure: Count of Participants; unit: Participants
Arm/Group | IGRT/VMAT Focal Therapy Boost to DIL
Number analyzed (Participants) | 30
Participants | 30

5. Secondary Outcome: Quality of Life (QoL) Assessed by the Expanded Prostate Cancer Index Composite EPIC16 Scale 0-60 (Best to Worst). The Total Score of the Scale is the Summatory of the Domain's Score
Description: Assessment of the QoL perceived by the patient in the urinary incontinence, urinary abstraction irritation, bowel function, sexual function and vitality/hormone functions domains
Time Frame: 5 years
Population: No clinical data were collected for this outcome.
Arm/Group | IGRT/VMAT Focal Therapy Boost to DIL
Number analyzed (Participants) | 0

6. Secondary Outcome: Disease-free Survival (DFS)
Description: Survival free of any event including biochemical failure, local failure, distant metastasis or death
Time Frame: 5 years
Reporting Status: Not Posted

7. Secondary Outcome: Verification of Safety Margins
Description: Quantification of the systematic and random errors during the preparation and administration of the radiotherapy treatment in 15 patients. Security margins estimation according to Van Herk formula
Time Frame: 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | IGRT/VMAT Focal Therapy Boost to DIL
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 27/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IGRT/VMAT Focal Therapy Boost to DIL (N=30)
Acute rectal toxicity (Gastrointestinal disorders) | 2 (2)
Acute urinary toxicity (Renal and urinary disorders) | 19 (19)
Late rectal toxicity (Gastrointestinal disorders) | 3 (3)
Late urinary toxicity (Renal and urinary disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-18): https://cdn.clinicaltrials.gov/large-docs/25/NCT03030625/Prot_SAP_000.pdf